CLINICAL TRIAL: NCT03198689
Title: A Pilot Study of Adcetris Treatment in Active Diffuse Cutaneous Systemic Sclerosis (Diffuse Scleroderma)
Brief Title: Brentuximab Vedotin in Early Diffuse Cutaneous Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Principal Investigator, Janet Pope, Head of Rheumatology, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BV201708
Record Dates: First submitted 2017-06-14; First posted 2017-06-26 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis
Keywords: systemic sclerosis; scleroderma; brentuximab vedotin; CD30-directed antibody-drug conjugate; antirheumatic agents; antineoplastic agents; connective tissue diseases; skin diseases; immunologic factors
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic; Connective Tissue Diseases; Skin Diseases | interventions — Brentuximab Vedotin

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Administration of Brentuximab vedotin (Experimental): Maximum duration of treatment: 48 weeks Maximum dose allowed: 0.6 mg/kg Route of administration: intravenous use
  Interventions: Drug: Brentuximab Vedotin

INTERVENTIONS:
Drug: Brentuximab Vedotin — Dose 0.6 mg/kg i.v. will be given every 3 weeks for 16 cycles (48 weeks) in addition to standard of care medications for SSc that may include cyclophosphamide, methotrexate, azathioprine, mycophenylate mofetil (MMF, cellcept) and mycophenolic acid (myfortic).
  Other Names: ADCETRIS, SGN-35

SUMMARY:
The purpose of this study is to assess feasibility, safety and preliminary efficacy of Brentuximab vedotin (Adcetris), a CD30-directed antibody-drug conjugate, in the treatment of active diffuse cutaneous systemic sclerosis (dcSSc).

DETAILED DESCRIPTION:
Systemic sclerosis (SSc, Scleroderma) is a multisystem autoimmune disease characterized by widespread vascular injury and progressive fibrosis of the skin and internal organs. Internal organ involvement results in increased mortality of SSc patients. There is no effective treatment for the majority of patients with early active diffuse scleroderma (diffuse cutaneous systemic sclerosis; dcSSc). These patients early in their disease may be able to reverse their inflammation and reduce the probability of irreversible fibrosis via significant immune modulation. This is a pilot study that will treat 10 patients with early or active dcSSc who meet inclusion criteria to determine if the benefit of Brentuximab vedotin and safety are favorable in order to consider a randomized controlled trial. This is a Phase II study that is uncontrolled and patients will remain on their background immune suppressive treatment unless if contraindicated for safety or drug interactions. The trial is powered to show a mean change in mRSS of 8 over one year in an uncontrolled, unblinded study. The Health Assessment Questionnaire Disability Index (HAQ), patient and physician global scores, inflammatory markers (ESR, CRP), and combined response index in SSc (CRISS) will all be exploratory outcomes. Other outcomes such as changes in CD30-stained cells on skin biopsies with IHC from baseline to end of the trial will be explored if the study is positive.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* able to give informed consent
* meet the ACR/EULAR classification criteria for SSc
* early dcSSc (disease duration ≤ 5 years from first non-Raynaud's phenomenon symptom) OR active dcSSc as determined by worsening mRSS, presence of tendon friction rubs, and/or elevated inflammatory markers thought to be due to active dcSSc and not related to other issues
* mRSS≥ 15
* a negative TB skin test at screening, or treatment with INH for 6 months or other standardized LBTI (latent TB infection) treatment in the past

Exclusion Criteria:

1. Poor pulmonary function (FVC<40% and/or DLCO<30%).
2. Pregnancy, breast feeding or child bearing potential without practicing reliable contraception (and partners for men in the study).
3. Clinically significant pulmonary hypertension requiring drug therapy.
4. Clinically significant cardiac disease.
5. Chronic or ongoing active infectious disease requiring systemic treatment.
6. Seropositivity for human immunodeficiency virus (HIV) at study entry.
7. Active tuberculosis (TB) infection.
8. Active viral infection with viral replication of hepatitis B or C virus at study entry.
9. Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, pancreatic, haematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease; and cancer.
10. Peripheral neuropathy at screening Grade 2 or higher.
11. Known or suspected hypersensitivity to components of the treatment
12. Patients known or suspected of not being able to comply with a study protocol (e.g. due to alcoholism, drug dependency or psychological disorder)
13. Any of the following laboratory abnormalities at screening:

    * Absolute neutrophils count <2000/mm3
    * Hemoglobin <85 g/L
    * Platelet count < 100,000/mm3
    * AST/SGOT or ALT/SGPT >2.0 UNL
14. Participation in another clinical trial within six weeks before randomization in this study
15. Use of rituximab within the previous 4 months.
16. Immunization with a live/ attenuated vaccine less than 4 weeks prior to the baseline visit.
17. Previous use of brentuximab vedotin.
18. Current or history of progressive multifocal leukoencephalopathy (PML).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Change in skin thickness measured by modified Rodnan Skin Score (mRSS) | 12 months

SECONDARY OUTCOMES:
Change in mRSS | 3, 6 and 9 months
CRISS score >20% | 6 months
Change in FVC, % | 6 and 12 months
Change in DLCO, % | 6 and 12 months
Change in physician-assessed disease activity, severity and damage on VASs ranked from 0 to 10 | 3,6,9 and 12 months
Change in patient global assessment of health status (VAS 0 to 10) | 3,6,9 and 12 months
Change in Health Transition score | 3,6,9 and 12 months
Change in SHAQ | 3,6,9 and 12 months

OTHER OUTCOMES:
Change in blood levels of soluble CD30 | 3,6,9 and 12 months
Change in serum levels of sIL-2R | 3,6,9 and 12 months
Change in serum levels of aminoterminal propeptide of type III collagen | 3,6,9 and 12 months
Change in myofibroblast score in skin biopsies of involved forearm skin | 6 and 12 months
Change in CD30-positive cell count in skin biopsies of involved forearm skin | 6 and 12 months
Change in erythrocyte sedimentation rate | 3,6,9 and 12 months
Change in hsCRP levels | 3,6,9 and 12 months
Number of patients with infectious complications | up to 1 month post-treatment
Number of patients with regimen-related toxicities | up to 12 weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Janet E Pope, Principal Investigator — University of Western Ontario, Division of Rheumatology, St. Joseph's Health Care, London, Ontario, Canada
Locations (1):
- Rheumatology Clinic, St. Joseph's Health Care, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Young A, Khanna D. Systemic sclerosis: a systematic review on therapeutic management from 2011 to 2014. Curr Opin Rheumatol. 2015 May;27(3):241-8. doi: 10.1097/BOR.0000000000000172. PMID 25775190
- [Background] Shah AA, Casciola-Rosen L, Rosen A. Review: cancer-induced autoimmunity in the rheumatic diseases. Arthritis Rheumatol. 2015 Feb;67(2):317-26. doi: 10.1002/art.38928. No abstract available. PMID 25371098
- [Background] Pope JE, Baron M, Bellamy N, Campbell J, Carette S, Chalmers I, Dales P, Hanly J, Kaminska EA, Lee P, et al. Variability of skin scores and clinical measurements in scleroderma. J Rheumatol. 1995 Jul;22(7):1271-6. PMID 7562757
- [Background] Furst DE, Khanna D, Mattucci-Cerinic M, Silman AJ, Merkel PA, Foeldvari I; OMERACT 7 Special Interest Group. Scleroderma--developing measures of response. J Rheumatol. 2005 Dec;32(12):2477-80. PMID 16331791
- [Background] Pope JE, Bellamy N. Outcome measurement in scleroderma clinical trials. Semin Arthritis Rheum. 1993 Aug;23(1):22-33. doi: 10.1016/s0049-0172(05)80024-1. PMID 8235663
- [Background] Sutherland MS, Sanderson RJ, Gordon KA, Andreyka J, Cerveny CG, Yu C, Lewis TS, Meyer DL, Zabinski RF, Doronina SO, Senter PD, Law CL, Wahl AF. Lysosomal trafficking and cysteine protease metabolism confer target-specific cytotoxicity by peptide-linked anti-CD30-auristatin conjugates. J Biol Chem. 2006 Apr 14;281(15):10540-7. doi: 10.1074/jbc.M510026200. Epub 2006 Feb 16. PMID 16484228
- [Derived] Fernandez-Codina A, Nevskaya T, Baron M, Appleton CT, Cecchini MJ, Philip A, El-Shimy M, Vanderhoek L, Pinal-Fernandez I, Pope JE. Brentuximab vedotin for skin involvement in refractory diffuse cutaneous systemic sclerosis, an open-label trial. Rheumatology (Oxford). 2025 Mar 1;64(3):1476-1481. doi: 10.1093/rheumatology/keae235. PMID 38652570